CLINICAL TRIAL: NCT01013415
Title: A Phase I/II Study Of the Safety, Survival, and Trafficking of Autologous CD4-ZETA Gene-Modified T Cells With and Without Extension Interleukin-2 in HIV Infected Patients
Brief Title: CD4-ZETA Gene Modified T Cells With and Without Exogenous Interleukin-2 (IL-2) In HIV Patients
Acronym: CD4-ZETA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WU #8829-99
Record Dates: First submitted 2009-11-05; First posted 2009-11-13 (Estimated); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: HIV-1 Infections
Keywords: HIV-1
MeSH Terms: interventions — Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ARM 1 (Experimental): Arm I (N=5) received antiretroviral therapy (ART) plus low dose IL-2 (1.2 million units/m2) subcutaneously daily for 56 days
  Interventions: Drug: HAART
- ARM 2 (Experimental): Arm 2 (N=5) received ART plus a single infusion of approximately 5 to 11 billion CD4-zeta gene modified T cells.
  Interventions: Biological: T cells
- ARM 3 (Experimental): Arm 3 (n=5) received ART plus IL-2 (1.2 million units/m2) and a single infusion of approximately 5 to 11 billion CD4-zeta gene modified T cells.
  Interventions: Drug: HAART; Biological: T cells

INTERVENTIONS:
Drug: HAART
  Other Names: ARM 1, ARM 2, ARM 3
  Arms: ARM 1; ARM 3
Biological: T cells
  Other Names: ARM 2, ARM 3
  Arms: ARM 2; ARM 3

SUMMARY:
The purpose of this study is to find out the safety and activity of an experimental anti-HIV treatment using autologous CD4-zeta gene-changed T cells and/or IL-2 (recombinant interleukin2).

DETAILED DESCRIPTION:
The purpose of this study is to find out the safety and activity of an experimental anti-HIV treatment using autologous CD4-zeta gene-changed T cells and/or IL-2 (recombinant interleukin2). The treatments that the investigators are studying try to improve the immune system by changing some of your T cells so they can find and destroy HIV infected cells (HIV is usually able to hide from your T cells). In this study, the investigators are also trying to find out if giving you more IL-2 at the same time as gene changed T cells will help the T cells to live longer or fight HIV better.

ELIGIBILITY:
Inclusion Criteria:

* DOD beneficiary with HIV-1 infection
* Greater than or equal to 200 CD4 cells/mm3
* Undetectable viral load, for at least the previous 8 weeks
* Stable anti-retroviral regimen for greater than or equal to 8 weeks
* Venous access sufficient for apheresis
* Karnofsky performance > 80%

Exclusion Criteria:

* Inadequate organ function
* Lifetime history of CD4 count less than 200 cells/mm3 on 2 consecutive measurements over at least an 8 week period
* Any previous history of gene therapy
* Recent IL-2 therapy or other treatment with an investigational agent
* Pregnancy
* some medications (hydroxyurea, corticosteroids and other immunosuppressants, chemotherapy, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2001-09; Primary Completion 2005-06 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Safety of CD4-zeta T cells with and without IL-2 in the setting of HAART | Through study completion, an average of 1 year
  To assess and compare the safety of each arm when comparing related adverse events reported of subjects on study through the end of study (week 54).
Effect of IL-2 on the Persistence of CD4-zeta T cells | Through study completion, an average of 1 year
  Subjects who received IL-2 plus gene-modified cells versus those who received cells alone will have greater numbers gene-modified cells in both PBMCs and rectal lymphoid tissue. This will be done by quantifying residual virus in the reservoir using more modern techniques that permit quantification of small amounts of virus in the rectal lymphoid tissue and to quantify specifically replication competent HIV (versus total HIV).
To compare the viral load of subjects from baseline to the end of study. | Through study completion, an average of 1 year
  Determine the effect of CD4-zeta infusions with and without IL-2 on viral load (plasma HIV-1 RNA, tissue HIV-1 RNA, and frequency of latent replication-competent HIV-1 in PBMC) at study specific timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Aronson, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No